CLINICAL TRIAL: NCT01084902
Title: Comparison of the Effects of Latanoprost(0.005%) and Brinzolamide(1.0%) on Intraocular Pressure in Primary Open-angle Glaucoma and Ocular Hypertension
Brief Title: Efficacy Comparison of Xalatan and Azopt on POAG and OH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Yingzi PAN/Professor of Ophthalmological Department, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKU1H001; PKU1H (Other Grant/Funding Number: IIR)
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Last update posted 2010-03-11 (Estimated); Status verified 2010-03

CONDITIONS: Ocular Hypertension
Keywords: POAG; OH; Xalatan; Azopt; Primary Open Angle Study
MeSH Terms: conditions — Ocular Hypertension | interventions — Latanoprost; brinzolamide

ARMS (2):
- latnoprost (Experimental): once daily
  Interventions: Drug: Latanoprost
- Brinzolamide (Active Comparator): two times daily
  Interventions: Drug: Brinzolamide

INTERVENTIONS:
Drug: Latanoprost — once daily
  Arms: latnoprost
Drug: Brinzolamide — Two times daily
  Arms: Brinzolamide

SUMMARY:
Prostaglandin analogs (PGAs) represent a new class of active ocular hypotensive agents and possess a unique mechanism of action. Many studies suggested that 0.005% Latanoprost was more effective and safer than other anti-glaucoma medications, such as beta-blockers. It has also been found to be more effective than other class of anti-glaucoma medications such as carbonic anhydrase inhibitors and alpha agonists. However data on such comparison is lacking in Chinese patients. So it is necessary to increase China experience and get clinical data from China. Besides latanoprost, brinzolamide is known as one of the other ocular hypotensive agents with less systemic adverse effects, therefore it is selected as the controlled medication of this study. The administration phase will be 4 weeks because it is long enough to compare both efficacy and safety of the study drugs and accounting for following-up conditions in China, it will be easier for the investigators to get enough subjects in a limited stage if the observation time is shorter.

Before treatment with the study drugs, any previous glaucoma drugs will be washed out. The minimum washout periods are 5 days for cholinergic agonists, 1 week for adrenergic agonists, 3 weeks for adrenergic β receptor blockers and 4 weeks for PGAS. After washout, the patients will be randomised send to two parallel study groups: one group will receive latanoprost 0.005% once daily in the evening, the other group receive 1.0% Brinzolamide twice daily. Randomization will be obtained using a list of random numbers .During the study there will be four visits: screening, baseline, 2 weeks, and 4 weeks of treatment. The IOP will be measured with a Goldmann tonometer at 8 am for each visit. The tonometry will be performed before the administration of the dose of the day in patients treated with Brinzolamide. Three separate measurements will be taken for each eye and the mean of the three measurements will be used in the statistical analysis. Best corrected visual acuity and refraction will be determined and a slit lamp examination, ophthalmoscopy will be performed at all visits.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with POAG or OHT
2. Older than 18 years, either sex
3. With IOP≤30mmHg in both eyes and with IOP>21mmHg in either eye after washout
4. Understand the study instructions and are willing to attend at all follow-up appointments
5. Be willing to comply with study medication use
6. Ready for written informed consent

Exclusion Criteria:

1. Visual field defects within the central 10°
2. Absence of vision in one eye
3. History of hypersensitivity to any components of the study medications
4. Contraindications to carbonic anhydrase inhibitors or prostaglandins
5. History of ocular herpetic disease, uveitis, or cystoid macular edema
6. Ocular history of trauma, inflammation, surgery or use of corticosteroids (within 2 months)
7. History of ocular laser therapy within 3 months
8. Severe dry eyes
9. Signs of ocular infection, except blepharitis
10. Corneal abnormality that may affect IOP measurements
11. Unwilling to accept the risk for hyperchromia of the iris or development of hypertrichosis
12. Pregnant females or lactating mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2010-02; Primary Completion 2010-09 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Intraocular Pressure | Baseline, 2 weeks, 4 weeks
  Three separate measurements will be taken for each eye. And mean result will be taken if the difference between measurements is within 2 mmHg , or use the median if the difference between measurements is greater than 3 mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Yingzi Pan, doctor, Study Chair — Peking University First Hospital